CLINICAL TRIAL: NCT00169910
Title: VIP: Vascular Imaging Project. Prospective Randomized Study on the Effect of AUC-monitored Treatment With Steroids Combined With Either a Calcineurin Inhibitor or Mycophenolate Mofetil on the Progression of Subclinical Cardiovascular Disease in Renal Transplant Recipients.
Brief Title: VIP: Vascular Imaging Project. Study on the Progression of Cardiovascular Disease in Renal Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, J.S.Mourer, MD, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P05.105
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Cardiovascular Disease
Keywords: Renal Transplantation; Calcineurin Inhibitor; Mycophenolate Mofetil; Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — cni protein, Drosophila

ARMS (2):
- 1 (Active Comparator): AUC monitored withdrawal of MMF
  Interventions: Drug: AUC monitored withdrawal of MMF or CNI
- 2 (Active Comparator): AUC monitored withdrawal of CNI
  Interventions: Drug: AUC monitored withdrawal of MMF or CNI

INTERVENTIONS:
Drug: AUC monitored withdrawal of MMF or CNI — AUC monitored withdrawal of MMF or CNI from a immunosuppressive drug regimen with steroids, CNI and MMF in stable renal transplant recipients

SUMMARY:
This is a prospective randomized study to compare the influence of area under the curve (AUC)-monitored dual treatment with steroids in combination with either a calcineurin inhibitor (CNI) or mycophenolate mofetil (MMF) on the progression of subclinical cardiovascular disease in renal transplant recipients.

Since CNI have a detrimental effect on cardiovascular risk factors, it is the researchers' hypothesis that renal recipients after CNI withdrawal will have more reduction of markers of cardiovascular disease.

DETAILED DESCRIPTION:
Stable renal transplant patients on maintenance immunosuppressive therapy with steroids, a calcineurin inhibitor (CNI) and mycophenolate mofetil (MMF) will be randomized for AUC-monitored withdrawal of either CNI or MMF.

The progression of cardiovascular markers will be assessed by yearly measurements of Intima Media Thickness, Pulse Wave Velocity and Left Ventricular Hypertrophy in both groups.

The duration of the study will be 3 years and the target sample size is 100 patients per arm

ELIGIBILITY:
Inclusion Criteria:

* Patients, 18 years or older, on triple maintenance therapy with cyclosporine or tacrolimus , MMF and steroids
* Informed consent

Exclusion Criteria:

* Calculated creatinine clearance < 30 ml/min
* Multi-organ recipients
* Patients with a (historic) panel reactive antibody (PRA) >60%
* Third renal transplant or more.
* Patients receiving investigational drugs other than MMF in combination with cyclosporine or tacrolimus
* Solid malignancy, post-transplant lymphoproliferative disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2005-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Primary endpoint: progression of subclinical cardiovascular disease as assessed by intima media thickness (IMT), pulse wave velocity (PWV) and left ventricular hypertrophy (LVH) | 3 years

SECONDARY OUTCOMES:
Secondary endpoint: Cardiovascular risk factors: a) Hypertension, b) Hyperlipidemia, c) Diabetes mellitus/glucose intolerance | 3 years
Graft function | 1 year, 3 years
Incidence of acute rejection | 1 year, 3 years
Graft survival (creatinine clearance < 15 ml/min or dialysis) | 1 year, 3 years
Patient survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Johan W. de Fijter, MD,PhD, Study Chair — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

REFERENCES:
- [Background] Schnuelle P, van der Heide JH, Tegzess A, Verburgh CA, Paul LC, van der Woude FJ, de Fijter JW. Open randomized trial comparing early withdrawal of either cyclosporine or mycophenolate mofetil in stable renal transplant recipients initially treated with a triple drug regimen. J Am Soc Nephrol. 2002 Feb;13(2):536-543. doi: 10.1681/ASN.V132536. PMID 11805185
- [Background] O'Leary DH, Polak JF, Kronmal RA, Manolio TA, Burke GL, Wolfson SK Jr. Carotid-artery intima and media thickness as a risk factor for myocardial infarction and stroke in older adults. Cardiovascular Health Study Collaborative Research Group. N Engl J Med. 1999 Jan 7;340(1):14-22. doi: 10.1056/NEJM199901073400103. PMID 9878640
- [Background] Blacher J, Guerin AP, Pannier B, Marchais SJ, Safar ME, London GM. Impact of aortic stiffness on survival in end-stage renal disease. Circulation. 1999 May 11;99(18):2434-9. doi: 10.1161/01.cir.99.18.2434. PMID 10318666
- [Derived] Mourer JS, de Koning EJ, van Zwet EW, Mallat MJ, Rabelink TJ, de Fijter JW. Impact of late calcineurin inhibitor withdrawal on ambulatory blood pressure and carotid intima media thickness in renal transplant recipients. Transplantation. 2013 Jul 15;96(1):49-57. doi: 10.1097/TP.0b013e3182958552. PMID 23715049